CLINICAL TRIAL: NCT05937698
Title: The CATALYST Study: Catalyzing Access to New Prevention Products to Stop HIV
Brief Title: The CATALYST Study
Status: Terminated | Type: Observational
Why Stopped: Study was stopped due to the stop work order issued by USAID on January 27, 2025.
Sponsor: FHI 360 (Other)
Collaborators: Wits Reproductive Health and HIV Institute (Other); LVCT Health (Other); Pangaea Zimbabwe Aids Trust (Other); Jhpiego (Other); United States Agency for International Development (USAID) (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: FHI 360 CATALYST
Record Dates: First submitted 2023-06-16; First posted 2023-07-10 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: HIV Prevention
Keywords: Pre-exposure prophylaxis (PrEP); oral PrEP containing tenofovir; dapivirine vaginal ring; injectable cabotegravir; adolescent girls and young women (AGYW)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood and/or dried blood spot
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The CATALYST study is an implementation study that will characterize and assess the implementation of an enhanced service delivery package providing informed choice of pre-exposure prophylaxis (PrEP) products among women at PEPFAR sites in Kenya, Lesotho, South Africa, Uganda, and Zimbabwe.

DETAILED DESCRIPTION:
The overall study goal is to characterize and assess the implementation of an enhanced service delivery package providing informed choice of pre-exposure prophylaxis (PrEP) products among women at U.S. President's Plan for AIDS Relief/U.S. Agency for International Development (PEPFAR/USAID) delivery sites in Kenya, Lesotho, South Africa, Uganda, and Zimbabwe. The study will be conducted in two stages, with currently approved oral PrEP and PrEP rings offered in Stage I, and the addition of CAB PrEP in Stage II after it has been approved by the regulatory authority in each country. The study goal will be accomplished by conducting a mixed-methods implementation study involving several components:

1. Component 1: Prospective cohort study of women at PEPFAR/USAID delivery sites that are delivering HIV PrEP, including daily oral PrEP, monthly PrEP rings, and bimonthly CAB PrEP

   1. Descriptive nested cohort study to evaluate the performance characteristics of different HIV testing strategies among participants who initiate CAB PrEP
   2. Descriptive nested cohort study to evaluate the feasibility and validity of a prevention effective use (PEU) measure among a subset of PrEP users
2. Component 2: Mixed-methods process evaluation involving implementers and key stakeholders

   1. Nested costing study across Lesotho, Uganda, and Zimbabwe study sites
   2. Nested qualitative study to understand community acceptance of PrEP and informed choice of PrEP products

ELIGIBILITY:
Inclusion Criteria:

* Tested HIV-negative as determined by the national HIV testing algorithm at a CATALYST site on the same day as enrollment
* Self-identify with at least one of the following populations:

  1. Adolescent girl or young women (AGYW) ages 15-24 years
  2. Female sex worker (FSW) ages 18 years and older
  3. Pregnant and breastfeeding populations (PBFP) ages 15 years and older
  4. Individuals assigned female at birth of any gender identity ages 15 years and older
  5. Individuals assigned male at birth who identify as women ages 15 years and older
  6. Other women ages 25 years and older
* Interested in learning about HIV prevention
* Willing to be contacted for follow-up by phone or other means (e.g., through a community health worker)
* Willing and able to provide informed written consent for participation

Exclusion Criteria:

* For participants ages 15-17 years, potential participants under the age of 18 may be excluded from study participation based on country guidelines and the age of consent. This determination will vary by country, including countries' definitions of emancipated minors. Country-specific informed consent forms will outline the country-specific inclusion criteria related to age.
* Certain sub-categories of participants may be excluded based on country guidelines.

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Individuals assigned female at birth of any gender identity or individuals assigned male at birth who identify as women are eligible to participate
Study Population: HIV-negative women* attending PEPFAR/USAID-supported facilities who are interested in learning about HIV prevention and are otherwise eligible to participate in the study
  *Presumed HIV-negative based on results from the national testing algorithm. For this study, the term "women" is inclusive of individuals assigned female at birth of any gender identity or individuals assigned male at birth who identify as women, although this definition is subject to local country guidelines.
Sampling Method: Non-Probability Sample
Enrollment: 6069 (Actual)
Dates: Start 2023-05-30 (Actual); Primary Completion 2025-01-27 (Actual); Study Completion 2025-01-27 (Actual)

PRIMARY OUTCOMES:
Overall and method-specific PrEP method uptake | 24 months
  Proportion of cohort members who initiate oral PrEP, the PrEP ring, CAB PrEP, or decline all PrEP or are ineligible for PrEP
Patterns of PrEP use | 24 months
  Person-time of continued use of a certain PrEP method, until switching to another method or missed resupply; Person-time of pause between missed resupply and reinitiation or switching (subset).
Qualitative assessment of health system feasibility | 24 months
  The extent to which PrEP choice and the enhanced service delivery package can be successfully carried out at facilities within health systems involved in CATALYST. This measure will be assessed through qualitative data collected through periodic in-depth interviews conducted among PrEP providers, community stakeholders, and key informants at selected sites.
Delivery acceptability among providers measured using an adapted version of the Acceptability of Intervention Measure (AIM) | 24 months
  Perception that offering informed choice of PrEP products and the provision of the enhanced service delivery package are agreeable or satisfactory in this setting as measured though an adapted version of the acceptability of intervention measure (Weiner et al. 2017), a 5-item scale with higher scores representing greater acceptability (range: 5-25).

OTHER OUTCOMES:
Cost of delivery at a subset of study sites | 24 months
  The cost of the implementation effort, including average unit cost estimates for oral PrEP, the PrEP ring, and CAB PrEP in Lesotho, Uganda, and Zimbabwe and the incremental unit cost of adding PrEP ring and CAB PrEP at sites already providing oral PrEP
Qualitative assessment of community acceptability of PrEP and PrEP choice | 24 months
  Perception that PrEP (and PrEP choice) are agreeable, satisfactory, and welcomed in the community, especially among primary PrEP influencers (partners and parents/caregivers). This measure will be assessed through qualitative in-depth interviews conducted among primary PrEP influencers in select CATALYST communities, including parents/caregivers of existing and potential PrEP users and partners of existing and potential PreP users.
Product acceptability among users as assessed through a theory-informed questionnaire relating to different aspects of acceptability (Sekhon et al., 2022) | 24 months
  Perception that PrEP product is agreeable or satisfactory. This measure will be assessed through administration of an adapted version of the theory-informed questionnaire developed by Sekhon et al., 2022. Item scores will be reported separately for each acceptability construct.
Prevention effective use of PrEP products | 24 months
  Percent of risk-days (days with condomless sex) when participants were protected from HIV acquisition by taking PrEP based on reported daily occurrence within certain periods. Note that this measure will only be reported if measure passes validation assessment conducted early in the implementation period.
Rates of HIV infection among participants | 24 months
  Number of study cohort members who become infected with HIV at any point during the study disaggregated by PrEP use status after enrollment (but not including the enrollment visit).
Rates of HIV drug resistance among PrEP users who acquire HIV during study participation | 24 months
  Number and type of HIV drug resistance-associated polymorphisms and/or mutations identified among participants who become infected with HIV and were exposed to PrEP
Pregnancy and selected infant outcomes among pregnant and breastfeeding populations for outcomes occurring during the study period. | 24 months
  Among pregnant participants reporting exposure to PrEP during pregnancy: type and frequency of pregnancy outcomes (term live birth [≥37 weeks], preterm live birth [<37 weeks], pre-term birth, stillbirth, birth weight and sex, spontaneous abortion, congenital anomalies, gestational age, neonatal death) among outcomes occurring during the study period
Frequency of reported side effects by PrEP product | 24 months
  The type, number, and perceived severity of patient-reported side effects from PrEP product use

CONTACTS AND LOCATIONS:
Overall Officials: Virginia Fonner, Study Chair — FHI 360; Elizabeth Irungu, Study Chair — Jphiego; Kevin K'Orimba, Principal Investigator — LVCT Health; Nicolette Naidoo, Principal Investigator — Wits RHI; Carolyne Akello, Principal Investigator — FHI 360 Uganda; Emily Gwavava, Principal Investigator — Pangaea Zimbabwe Aids Trust
Locations (28):
- Kenya (6):
  - Chulaimbo sub-country hospital, Kisumu
  - Migosi Health, Kisumu
  - Likoni Sub-country hospital, Mombasa
  - Tudor sub-country hospital, Mombasa
  - Bar Hostess Empowerment & Support Programme (BHESP) Drop-In Centre, Nairobi
  - Mukuru Public Health Centre, Nairobi
- Lesotho (3):
  - Sefika, Maseru
  - Scott Hospital, Morija
  - Berea, Teyateyaneng
- South Africa (6):
  - Phomolong Clinic, Hennenman
  - FSW Esselen Street, Johannesburg
  - TG Esselen Street, Johannesburg
  - Hani Park Clinic, Welkom
  - Matjhabeng Clinic, Welkom
  - Welkom Clinic, Welkom
- Uganda (7):
  - Gulu RRH, Gulu
  - Bufunda HC III, Ibanda
  - Kitgum Hospital, Kitgum
  - Namakwekwe HC III, Mbale
  - Mbarara HC IV, Mbarara
  - Bison HCCIII, Tororo
  - Malaba HC III, Tororo
- Zimbabwe (6):
  - Beitbridge Wellness Clinic, Beitbridge
  - Cowdray Park Clinic, Bulawayo
  - Plumtree District Hospital, Bulawayo
  - SHAZ! Hub (Citimed Hopstial), Chitungwiza
  - Runyararo Clinic, Masvingo
  - Ngundu Rural Health Center, Ngundu

IPD SHARING:
Plan to Share IPD: Yes
In accordance with the USAID Automated Directives System 579, after acceptance of any knowledge product presenting study findings and after being cleaned of any information that could be used to personally identify participants, the quantitative survey dataset along with relevant documentation will be registered with USAID's Development Data Library (DDL) and made publicly available in an open data repository, to the extent permissible by participating countries' privacy and data sharing regulations.
Supporting Information: Study Protocol, ICF
Time Frame: After study completion and manuscript submission.

REFERENCES:
- See also: PrEP Watch: CATALYST — http://www.prepwatch.org/catalyst/